CLINICAL TRIAL: NCT00563147
Title: A Phase 1b, Open-Label, Dose-Finding Study to Evaluate the Safety of Tivozanib (AV-951) in Combination With Temsirolimus in Subjects With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-07-102
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Renal Cell Carcinoma
Keywords: tivozanib; AV-951
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tivozanib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): tivozanib (AV-951) plus temsirolimus
  Interventions: Drug: tivozanib (AV-951) plus temsirolimus

INTERVENTIONS:
Drug: tivozanib (AV-951) plus temsirolimus — ascending doses of tivozanib (AV-951) capsules administered orally for 21 days with discontinuation for 7 days; ascending doses of temsirolimus administered intravenously every 7 days
  Other Names: Torisel (temsirolimus)

SUMMARY:
The purpose of this study is to test the safety and tolerability of tivozanib (AV-951) and Torisel™ given in combination for renal cell cancer. The study will also assess the effects of the combination of tivozanib (AV-951) and Torisel™ on the tumor. Tivozanib (AV-951) is a VEGF-receptor tyrosine kinase inhibitor, and may stop the growth of tumor cells by blocking blood flow to the tumor. Temsirolimus is an mTOR inhibitor which is approved for the treatment of advanced renal cell carcinoma.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, dose-finding study of tivozanib (AV-951) in combination with temsirolimus to include approximately 36 subjects with metastatic renal cell carcinoma (mRCC). This study is designed to evaluate the safety, tolerability, dose-limiting toxicities (DLT), maximum tolerated dose (MTD), pharmacokinetic, pharmacogenomic, and antineoplastic activity of tivozanib (AV-951) when administered in combination with temsirolimus. Tivozanib (AV-951) will be administered once daily for 3 weeks beginning on Day 1 of Cycle 1, followed by 1 week off (1 cycle = 4 weeks). Temsirolimus will be administered intravenously once weekly starting on Day 8 of Cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18-year-old males or females
* Histologically confirmed renal cell carcinoma with a clear cell component
* Documented progressive disease
* Measurable disease by RECIST criteria
* No more than 1 prior VEGF receptor targeted therapy; no prior treatment with temsirolimus or other drugs targeting the mTOR pathway
* Karnofsky performance status > 70%; life expectancy ≥ 3 months
* Ability to give written informed consent

Exclusion Criteria:

* Known hypersensitivity to temsirolimus or its metabolites (including sirolimus), polysorbate 80, or to any other component of the temsirolimus formulation
* Primary CNS malignancies; active CNS metastases
* Hematologic malignancies (including leukemia in any form, lymphoma, and multiple myeloma)
* Any of the following hematologic abnormalities:

  * Hemoglobin < 9.0 g/dL
  * ANC < 1500 per mm3
  * Platelet count < 100,000 per mm3
* Any of the following serum chemistry abnormalities:

  * Fasting serum cholesterol > 350 mg/dL
  * Fasting triglycerides > 400 mg/dL
  * Total bilirubin > 1.5 × ULN
  * AST or ALT > 2.5 × ULN (or > 5 x ULN in subjects with liver metastasis)
  * Serum albumin < 3.0 g/dL
  * Creatine > 1.5 × ULN (or calculated CLCR <50 mL/min/1.73 m2)
  * Proteinuria > 2.5 g/24 hours or 3+ with urine dipstick
* Significant cardiovascular disease, including:

  * Active clinically symptomatic left ventricular failure
  * Active hypertension (diastolic blood pressure > 100 mmHg). Subjects with a history of hypertension must have been on stable doses of anti-hypertensive drugs for ≥ 4 weeks
  * Uncontrolled hypertension: Blood pressure >140/90 mmHg on 2 or more antihypertensive medications
  * Myocardial infarction within 3 months prior to administration of first dose of study drug
* Subjects with delayed healing of wounds, ulcers, and/or bone fractures
* Pulmonary hypertension or pneumonitis
* Serious/active infection; infection requiring parenteral antibiotics
* Inadequate recovery from any prior surgical procedure; major surgical procedure within 6 weeks prior to study entry
* Uncontrolled psychiatric disorder, altered mental status precluding informed consent or necessary testing
* Inability to comply with protocol requirements
* Ongoing hemoptysis or history of clinically significant bleeding
* Cerebrovascular accident within 12 months of study entry, or peripheral vascular disease with claudication on walking less than 1 block
* Deep venous thrombosis or pulmonary embolus within 6 months of study entry and/or ongoing need for full-dose oral or parenteral anticoagulation
* Subjects with a "currently active" second primary malignancy other than non-melanoma skin cancers. Subjects are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy and are considered by their physician to be < 30% risk of relapse.
* Pregnant or lactating women
* Known concomitant genetic or acquired immune suppression disease such as HIV

Prohibited medications:

* VEGF receptor (VEGFR) targeted therapy within 4 weeks prior to and during study
* Other signal transduction inhibitors, monoclonal antibodies, etc., within 4 weeks prior to and during study
* Immunotherapy or biological response modifiers within 4 weeks prior to and during study
* Systemic hormonal therapy within 4 weeks prior to and during study, with the exception of:

  * Hormonal therapy for appetite stimulation or contraception
  * Nasal, ophthalmic, and topical glucocorticoid preparations
  * Oral replacement therapy for adrenal insufficiency
  * Low-dose maintenance steroid therapy for other conditions
* Herbal preparations/supplements (except for a daily multivitamin/mineral supplement not containing herbal components) within 2 weeks prior to or during study
* Any experimental therapy 4 weeks prior to and during study
* Radiotherapy:

  * At least 2 weeks since prior local radiation therapy (ie, involving <25% of bone marrow) at the time of study entry
  * At least 4 weeks since prior radiation therapy involving ≥ 25% of bone marrow
* Treatment with CYP3A4 inducers or inhibitors during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-11; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of tivozanib (AV-951) when given in combination with temsirolimus | 4 weeks (1 cycle)

SECONDARY OUTCOMES:
To characterize the pharmacokinetic profile of tivozanib (AV-951) and temsirolimus when administered in combination | 8 weeks (2 cycles)
To evaluate the antineoplastic activity of tivozanib (AV-951) and temsirolimus when administered in combination | 8 weeks (2 cycles)
To evaluate the effect of tivozanib (AV-951) and temsirolimus on global and targeted gene expression patterns | 8 weeks (2 cycles)
To determine the maximum tolerated dose (MTD) of tivozanib (AV-951) when administered in combination with temsirolimus | 4 weeks (1 cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Zhang, M.D., Study Director — AVEO Pharmaceuticals
Locations (5):
- United States (5):
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Stanford University, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - The Methodist Hospital Research Institute, Houston, Texas

REFERENCES:
- [Derived] Fishman MN, Srinivas S, Hauke RJ, Amato RJ, Esteves B, Cotreau MM, Strahs AL, Slichenmyer WJ, Bhargava P, Kabbinavar FF. Phase Ib study of tivozanib (AV-951) in combination with temsirolimus in patients with renal cell carcinoma. Eur J Cancer. 2013 Sep;49(13):2841-50. doi: 10.1016/j.ejca.2013.04.019. Epub 2013 May 28. PMID 23726267